CLINICAL TRIAL: NCT00921947
Title: A Phase II, Randomized, Open-Label Study to Evaluate the Comparative Safety and Immunogenicity of 1.0 µg Intramuscular (i.m.) and 2.0 µg Subcutaneous (s.c.) Dosing With VAX102 (M2e-flagellin) in Healthy Adults
Brief Title: Comparative Safety and Immunogenicity of 1.0 µg Intramuscular (i.m.) and 2.0 µg Subcutaneous (s.c.) Dosing With VAX102 (M2e-flagellin) Universal Influenza Vaccine in Healthy Adults
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: VaxInnate Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: VAX102-09
Record Dates: First submitted 2009-06-15; First posted 2009-06-17 (Estimated); Results first posted 2011-08-22 (Estimated); Last update posted 2011-08-24 (Estimated); Status verified 2011-08

CONDITIONS: Influenza
Keywords: influenza vaccine; M2e; Universal influenza vaccine
MeSH Terms: conditions — Influenza, Human | interventions — VAX102 vaccine

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- VAX102 IM (Experimental): VAX102 given as 1 µg intramuscular (i.m.)
  Interventions: Biological: VAX102
- VAX102 SC (Experimental): VAX102 given as a 2 µg subcutaneous (s.c.) dose
  Interventions: Biological: VAX102

INTERVENTIONS:
Biological: VAX102 — Universal M2e influenza vaccine
  Other Names: STF2.4xM2e

SUMMARY:
1. To assess the safety, reactogenicity, tolerability, and adverse events (AEs) of the VAX102 vaccine in a two dose regimen (Day 0 and Day 28) at the 1.0 µg dose level delivered i.m., or the 2.0 µg dose level delivered s.c. in a healthy adult population.
2. To assess the immunogenicity (anti-M2e serum antibody concentration) of the VAX102 vaccine in a two dose regimen (Day 0 and Day 28) at the 1.0 µg dose level delivered i.m., or the 2.0 µg dose level delivered s.c. as measured by an enzyme-linked immunosorbent assay (ELISA) in a healthy adult population.

ELIGIBILITY:
Inclusion Criteria:

* Adult men or women aged 18 to 49 years inclusive.
* Able and willing to provide written informed consent to participate.
* Healthy, as determined by medical history, physical examination, and vital signs.
* Willing to receive the unlicensed (VAX102) vaccine given as an i.m. or s.c. injection.
* Willing to provide multiple blood specimens collected by venipuncture.
* Females should avoid becoming pregnant during the course of the study
* Women of childbearing potential must have a negative urine pregnancy test within 24 hours preceding receipt of the first and preceding receipt of the second (booster) vaccination.
* Must exhibit comprehension of the study requirements; expressed availability for the required study period and expect to reside in the study area during the entire study period, and ability to attend scheduled visits.

Exclusion Criteria:

* Persons under 18 years old or 50 years or older.
* Persons with chronic illnesses such as cancer, diabetes, liver or kidney disease.
* Person currently pregnant, nursing mothers or planning a pregnancy within one month of vaccination.
* Persons who have had a prior serious reaction to influenza vaccine.
* Persons with a history of anaphylactic-type reaction to injected vaccines.
* Persons with a history of drug or chemical abuse in the year preceding the study.
* Persons who received an influenza vaccine for the current influenza season or those who plan to receive an influenza vaccine while participating in the study.
* Persons who received any other vaccine within one week prior to enrollment (may delay enrollment).
* Persons who have had a respiratory illness or illness with fever within three days of study enrollment (may delay enrollment).
* Persons currently participating in another research study involving any study medications (medicines or vaccines).

Ages: 18 Years to 49 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2009-06; Primary Completion 2009-07 (Actual); Study Completion 2009-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David N Taylor, MD, Study Director — VaxInnate Corporation
Locations (1):
- Jean Brown Research, Salt Lake City, Utah, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- VAX102 IM: Given as 1 µg intramuscular
- VAX102 SC: Given as 2 µg subcutaneous
Period: Day 0
Arm/Group | VAX102 IM | VAX102 SC
Started | 30 | 30
Completed | 30 | 30
Not Completed | 0 | 0
Period: Day 28
Arm/Group | VAX102 IM | VAX102 SC
Started | 28 (2 subjects were lost to follow-up and did not receive the 2nd vaccination of 1.0 ug i.m.) | 30
Completed | 28 | 30
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | VAX102 IM | VAX102 SC | Total
Number analyzed (Participants) | 30 | 30 | 60
Age Continuous [Mean (Standard Deviation); unit: years] | 27.3 (7.64) | 26.7 (8.74) | 27 (8.14)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 15 | 28
  Male | 17 | 15 | 32

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Local and Systemic Symptoms Post Vaccination 1 (Day 0)
Description: Solicited local and general symptoms experienced within 7 days after vaccination 1.
Time Frame: 0 to 7 days after vaccination
Population: The population analyzed included all participants receiving at least 1 dose of the vaccine.
Measure: Number; unit: participants
Arm/Group | VAX102 1.0 µg i.m. | VAX102 2.0 µg s.c.
Number analyzed (Participants) | 30 | 30
participants
  Redness | 0 | 13
  Swelling | 2 | 3
  Bruising | 0 | 0
  Arm Pain | 23 | 21
  Headache | 5 | 3
  Fatigue | 4 | 4
  Joint Pain | 4 | 3
  Muscle Aches | 13 | 10
  Chills | 0 | 0
  Sweating | 1 | 1

2. Secondary Outcome: Anti-M2e Serum Antibody Concentration
Description: Anti-M2e Serum Antibody Concentration summarized by study visit using the per-protocol population.
Time Frame: 42 days (+/- 2)
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | VAX102 1.0 µg i.m. | VAX102 2.0 µg s.c.
Number analyzed (Participants) | 28 | 30
Titers
  Baseline | 0.011 [0.007 to 0.018] | 0.012 [0.008 to 0.019]
  Day 14 | 0.376 [0.206 to 0.685] | 0.375 [0.241 to 0.585]
  Day 28 | 0.255 [0.148 to 0.437] | 0.248 [0.165 to 0.374]
  Day 42 | 1.121 [0.744 to 1.689] | 2.062 [1.385 to 3.071]

3. Primary Outcome: Number of Participants With Local and Systemic Symptoms Post Vaccination 2 (Day 28)
Description: Solicited local and general symptoms experienced within 14 days after vaccination 2
Time Frame: 14 days after vaccination
Measure: Number; unit: participants
Arm/Group | VAX102 1.0 µg i.m. | VAX102 2.0 µg s.c.
Number analyzed (Participants) | 28 | 30
participants
  Redness | 0 | 0
  Swelling | 0 | 0
  Bruising | 0 | 0
  Arm pain | 0 | 0
  Headache | 0 | 0
  Fatigue | 0 | 1
  Joint Pain | 0 | 0
  Muscle Aches | 0 | 0
  Chills | 0 | 0
  Sweating | 0 | 0

ADVERSE EVENTS:
Time Frame: Serious adverse events were collected for 1 year following vaccination. All adverse events were collected for 42 days following vaccination.
Description: All reactogenicity findings were recorded in the CRFs. Symptoms from the Reactogenicity Memory Aid were reported as "reactogenicity", and presumed to be related to the investigational product. These complaints were not additionally recorded as AEs.
Arm/Group | VAX102 IM | VAX102 SC
Serious Adverse Events (participants affected / at risk) | 1/28 | 0/30
Other Adverse Events (participants affected / at risk) | 0/28 | 0/30
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | VAX102 IM (N=28) | VAX102 SC (N=30)
Hydronephrosis (Renal and urinary disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less